CLINICAL TRIAL: NCT05571514
Title: Study of the Impact of Mother-of-pearl Nutritional Supplementation on the Prevention of Post-menopausal Osteoporosis: Multicentre, Double-blind Randomized Versus Positive Comparator Study
Brief Title: Study of the Impact of Mother-of-pearl Nutritional Supplementation on the Prevention of Post-menopausal Osteoporosis
Acronym: NUTRANACRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20PH256; ANSM (Other: 2021-A01034-37)
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Post Menopausal Osteoporosis
Keywords: Mother-of-pearl; Osteoporosis; Ageing; Nutrition Health; Prevention
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Nacre; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: multicentre, double-blind randomized versus positive comparator study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stratified randomization :
  The study will be double-blinded to avoid follow-up bias and assessment bias. The maintenance of the blind will be guaranteed by the fact that the capsules of mother-of-pearl will be indistinguishable from those of CaCO3 (same shape, same color, same weight). Only the internal use pharmacies (IUP) of each center will be open, for the attribution of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother-of-pearl (Experimental): Patient randomized in the "Mother-of-pearl" group :
  Mother of pearl supplementation: 2 capsules of 400mg = 800mg mother of pearl/day, equivalent to 320mg Ca/day
  - Vitamin D: 50,000 IU/month (standard practice)
  Interventions: Dietary Supplement: Mother-of-pearl
- Calcium carbonate (Active Comparator): Patient randomized in the "Calcium carbonate" control group :
  Calcium carbonate supplementation: 2 capsules of 400mg= 800mg CaCO3/day, equivalent to 320mg Ca/day
  - Vitamin D: 50,000 IU/month (standard practice)
  Interventions: Dietary Supplement: Calcium Carbonate

INTERVENTIONS:
Dietary Supplement: Mother-of-pearl — The mother-of-pearl, derived from the inner shell of marine molluscs, is composed of calcium carbonate and organic compounds, some of which peptides are active on the bone.
  The mineralization inducing activity of the molecules extracted from the mother-of-pearl has been shown in vitro. Mother-of-pearl extract also contains molecules that inhibit the resorption activity of osteoclasts. Mother-of-pearl compounds can thus slow bone remodelling as showed in an ovariectomy-induced osteoporosis model in rat, where mother-of-pearl supplementation showed a better effect on limitation of bone loss than calcium carbonate supplementation.
  Arms: Mother-of-pearl
Dietary Supplement: Calcium Carbonate — Calcium carbonate is a source of calcium.
  Arms: Calcium carbonate

SUMMARY:
Post-menopausal osteoporosis and the resulting fractures are an important cause of disability and loss of independence. They also increase the risk of morbidity and mortality.

Given potential side effects, hormone replacement therapy is no longer recommended for menopausal women with risk of becoming osteoporotic. The very significant decrease in the use of these treatments is suspected of contributing to a resurgence in the incidence of osteoporotic fractures, particularly in women before the age of 70. There is a need for prevention of osteoporosis.

DETAILED DESCRIPTION:
Mother-of-pearl is a candidate for long-term use due to the combination of its effects: calcium supplementation, anti-resorptive activity and osteoanabolic activity.

Our hypothesis is that powdered mother-of-pearl supplementation limits bone loss in postmenopausal women with risk of becoming osteoporotic.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (50-65y) with risk of becoming osteoporotic
* T-score between -1 and -3
* Absence of fragility fractures history

Exclusion Criteria:

* absence of parathyroid glands (phospho-calcic regulation)
* presence of kidney stones
* patients who follow a treatment that could interfere with bone metabolism (corticotherapy, menopausal hormonal therapy, anti-oestrogen treatment, non-controlled hyperthyroiditis, hyper- and hypothyroiditis)
* bone diseases (Paget'disease, osteomalacia)
* chronic alcoholism

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in bone loss at lumbar site | Baseline from 12 months
  Demonstrate that oral mother-of-pearl powder supplementation, for 1 year, reduces bone loss at lumbar site in postmenopausal women with risk of becoming osteoporotic, in a better way than oral supplementation with pure CaCO3.
  Measurement of the change in BMD will be performed by DXA (dual X-ray absorptiometry bone densitometry)

SECONDARY OUTCOMES:
Tolerance to oral mother-of-pearl powder supplementation | Baseline from 12 months
  Tolerance will be assessed by collecting digestive disorders
Change in bone loss at the upper end of the femur | Baseline from 12 months
  Evaluate the impact of oral mother-of-pearl powder supplementation, compared to oral supplementation with pure CaCO3, for 1 year, in postmenopausal women on the bone loss at the upper end of the femur Measurement of the change in BMD will be performed by DXA (dual X-ray absorptiometry bone densitometry)
Change in bone remodeling of the femur | Baseline from 12 months
  Evaluate the impact of oral mother-of-pearl powder supplementation, compared to oral supplementation with pure CaCO3, for 1 year, in postmenopausal women on the bone remodeling Measurement of the change in BMD will be performed by measurement CTX (serum Collagen-telopeptide)

CONTACTS AND LOCATIONS:
Overall Officials: Adamah AMOUZOUGAN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (7):
- France (7):
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Clinique Universitaire de Rhumatologie, Grenoble
  - CH Emile Roux, Le Puy-en-Velay
  - Hôpital Edouard Herriot, Lyon
  - APHP - Hôpital Cochin, Paris
  - CH Roanne, Roanne
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No